CLINICAL TRIAL: NCT05812079
Title: Assessing the Protective Role of Insulin Like Growth Factor 1 Against Oxidative Stress in Vitiligo Patients
Brief Title: Insulin Like Growth Factor-1 Against Oxidative Stress in Vitiligo
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Salah El-Din El-Mesidy, Associate Professor, Cairo University
Other Study IDs: IGF-1 in Vitilgo
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: skin biopsy examined by ELISA technique — skin biopsy examined by ELISA technique

SUMMARY:
Insulin like growth factor has a protective role on melanocytes against the oxidative stress. The aim is to investigate this effect in vitiligo patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-segmental vitiligo

Exclusion Criteria:

1. Pregnant or lactating females
2. Smokers
3. Patients with any endocrinal disease known to affect GH or IGF-1 as Diabetes (by measuring HbA1c) and Thyroid disturbance (by measuring TSH)
4. Patients with liver disease (by measuring AST, ALT and GGT)
5. Obese patients (by measuring BMI)
6. Patients with history of ischemic heart disease (known medical history of angina or myocardial infarction or history of recurrent chest pain, left shoulder pain, shortness of breath or fatigue on the ordinary effort or less than the ordinary effort )
7. Patients with history of Peripheral arterial disease (Known medical history of peripheral arterial thrombosis or history of recurrent claudications)
8. Patients with history of cerebero-vascular disease (known medical history of transient ischemic attacks or stroke)
9. Patients who received systemic treatment for vitiligo during the previous six months or topical treatment during the previous two months

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Non-Segmental Vitiligo
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Investigate for IGF-1 and IMA levels in vitiligo | one year
  To measure the level of IGF-1 and the level of IMA in perilesional and distant skin of vitiligo patients and compare these levels with normal controls to investigate the relationship between IGF-1, as a protective from oxidative stress and IMA, as a marker of oxidative stress in vitiligo.

SECONDARY OUTCOMES:
Measure IMA in vitiligo and correlate it with psychological status of patients | One year
  To measure the serum level of IMA as a marker of oxidative stress in vitiligo patients versus normal controls 2- To correlate the findings with the VIS-22 score